CLINICAL TRIAL: NCT06277466
Title: Department of Pharmacy, the Affiliated Hospital of Xuzhou Medical University
Brief Title: Effect of Mutations in T2DM Susceptibility Genes on the Expression of Susceptibility Genes in Patients With T2DM and Controls
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: XYFY2023-KL478-01
Record Dates: First submitted 2024-02-05; First posted 2024-02-26 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Type 2 Diabetes Mellitus; Gene Polymorphisms; Genetic Mutations; Susceptibility, Genetic
Keywords: T2DM; gene polymorphism; susceptibility gene; genetic mutations
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Genetic Predisposition to Disease | interventions — Hypoglycemic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comparison of T2DM susceptibility gene expression between newly diagnosed T2DM patients and controls (Experimental): To determine the effect of gene mutations on the susceptibility of T2DM by comparing the expression levels of T2DM susceptibility genes in newly diagnosed T2DM patients and controls.
  Interventions: Drug: Fresh normal pancreatic tissues or adjacent tissues of pancreatic cancer were collected from controls and T2DM patients without hypoglycemic drugs; Drug: Fresh blood samples were collected from healthy subjects and T2DM patients without hypoglycemic drugs

INTERVENTIONS:
Drug: Fresh normal pancreatic tissues or adjacent tissues of pancreatic cancer were collected from controls and T2DM patients without hypoglycemic drugs — Compared with newly diagnosed T2DM patients, healthy subjects in the control group had normal levels of blood glucose, lipids, glycated hemoglobin levels, etc. Fresh normal pancreatic tissues or adjacent tissues of pancreatic cancer were collected before taking antidiabetic drugs in both groups.
Drug: Fresh blood samples were collected from healthy subjects and T2DM patients without hypoglycemic drugs — The newly diagnosed T2DM group should not have taken antidiabetic drugs and meet the diagnosis of T2DM. Fresh blood samples were collected before medication for detection.
  In the control group (healthy subjects), the indicators of physical examination were within the normal range and no hypoglycemic drugs were taken. Similarly, fresh blood samples should be taken for testing.

SUMMARY:
In this study, investigators wanted to determine the effect of T2DM susceptibility gene mutations on self-expression.

Participants (T2DM patients and controls) were recruited to identify genotypes and detect the levels of T2DM susceptibility genes expression in the fresh peripheral plasma. The normal pancreatic tissues or adjacent tissues of pancreatic cancer were also collected to identify the expression differences of T2DM susceptibility genes under different genotypes.

DETAILED DESCRIPTION:
The primary objective of this study was to investigate the changes of the expression of T2DM susceptible genes (NOS1AP, KCNQ1, TCF7L2, WSF1, GLP-1R, etc.) in participants (newly diagnosed T2DM patients and controls) after gene mutation.

Secondly, the expression differences of T2DM susceptible genes in T2DM patients with different genotypes were compared, and the relationship between the expression differences and clinicopathological characteristics of T2DM patients was analyzed.

Participants (newly diagnosed T2DM patients and healthy subjects) were screened from the department of endocrinology and health management center, whose fresh peripheral blood were collected. The normal pancreatic tissues or adjacent tissues of pancreatic cancer were collected in the department of general surgery. The DNA genome was extracted for genotyping, and then the expression levels of T2DM related susceptibility genes under different genotypes were detected by ELISA kits, PCR, WB,HE staining, IHC staining, ect.

The basic information of T2DM patients was collected, including demographic characteristics, physiological and biochemical data.Then investigators further compared the differences in the expression of susceptible genes between newly diagnosed T2DM patients and controls.

ELIGIBILITY:
Inclusion Criteria:

1. no drug therapy; 25 to 70 years old; Hemoglobin A1c (HbA1c) 7%-12%; BMI 20-35 kg/m2; Stable body weight (≤10% change within 3 months)（For newly diagnosed patients with T2DM）.
2. 25 to 60 years old; BMI 19-26 kg/m2; in good health, with no abnormalities of motor system, digestive system, respiratory system, urogenital system, blood system, circulatory system, nervous/mental system, endocrine system, etc（For healthy subjects）.
3. 20-80 years old; surgical resection of part or all of the pancreas; pancreatic lesions confirmed by enhanced CT or magnetic resonance (MR) examination or confirmed by intraoperative and postoperative pathology（For the patients in general surgical）.

Exclusion Criteria:

1. had taken antidiabetic drugs;
2. had a history of pancreatic surgery;
3. Complicated with severe organ lesions;
4. Long-term use of drugs that affect pancreatic function.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Detection of T2DM susceptibility gene expression in newly diagnosed T2DM patients | 1 month after fresh sample collection
  To detect the expression levels of susceptible genes in the plasma and the pancreatic tissues of newly diagnosed T2DM patients and compared with those in healthy subjects.
Detection of T2DM susceptibility gene expression in controls | 1 month after fresh sample collection
  To detect the expression levels of susceptible genes in the plasma and the pancreatic tissues of controls and compared with those in newly diagnosed T2DM patients.
Correlation between T2DM susceptibility gene expression and clinicopathological features | 6 months after obtaining the clinicopathological results
  Incidence of clinical pancreatic diseases under expression differences in T2DM susceptibility genes

SECONDARY OUTCOMES:
Baseline BMI of newly diagnosed with T2DM patients with different genotypes | 1 month of completion for individual screening
  Baseline BMI of newly diagnosed with T2DM patients
Baseline waist hip ratio (WHR) of newly diagnosed with T2DM patients with different genotypes | 1 month of completion for individual screening
  Baseline WHR of newly diagnosed with T2DM patients
Baseline fasting plasma glucose (FPG) of newly diagnosed with T2DM patients with different genotypes | 1 month of completion for individual screening
  Baseline FPG of newly diagnosed with T2DM patients
Baseline HbA1c of newly diagnosed with T2DM patients with different genotypes | 1 month of completion for individual screening
  Baseline HbA1c of newly diagnosed with T2DM patients
Baseline TC of newly diagnosed with T2DM patients with different genotypes | 1 month of completion for individual screening
  Baseline TC of newly diagnosed with T2DM patients
Baseline TG of newly diagnosed with T2DM patients with different genotypes | 1 month of completion for individual screening
  Baseline TG of newly diagnosed with T2DM patients
Baseline HDL-C of newly diagnosed with T2DM patients with different genotypes | 1 month of completion for individual screening
  Baseline HDL-C of newly diagnosed with T2DM patients
Baseline LDL-C of newly diagnosed with T2DM patients with different genotypes | 1 month of completion for individual screening
  Baseline LDL-C of newly diagnosed with T2DM patients
Baseline BMI of controls with different genotypes | 1 month of completion for individual screening
  Baseline BMI of controls
Baseline WHR of controls with different genotypes | 1 month of completion for individual screening
  Baseline WHR of controls
Baseline FPG of controls with different genotypes | 1 month of completion for individual screening
  Baseline FPG of controls
Baseline HbA1c of controls with different genotypes | 1 month of completion for individual screening
  Baseline HbA1c of controls
Baseline TC of controls with different genotypes | 1 month of completion for individual screening
  Baseline TC of controls
Baseline TG of controls with different genotypes | 1 month of completion for individual screening
  Baseline TG of controls
Baseline HDL-C of controls with different genotypes | 1 month of completion for individual screening
  Baseline HDL-C of controls
Baseline LDL-C of controls with different genotypes | 1 month of completion for individual screening
  Baseline LDL-C of controls

CONTACTS AND LOCATIONS:
Locations (1):
- China, Jiangsu, Department of Endocrinology, Xuzhou, China

IPD SHARING:
Plan to Share IPD: No